CLINICAL TRIAL: NCT07303348
Title: Multicenter Clinical Randomized Controlled Trial of Unilateral Biportal Endoscopic Spinal Surgery for Degenerative Grade 1 Spondylolisthesis Complicated With Lumbar Spinal Stenosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Changzheng Hospital (Other); Shanghai Kaiyuan Orthopedic Hospital (Unknown); Beijing Jishuitan Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Eastern Theater Command Naval Hospital (Unknown)
Responsible Party: Principal Investigator, Wei Xianzhao, Deputy Chief Physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPINE-UBE
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Spinal Stenosis (LSS); Degenerative Spondylolisthesis G1
Keywords: Grade Ⅰ degenerative spondylolisthesis; lumbar spinal stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perform surgery using the Unilateral Biportal Endoscopy (UBE) technique (Experimental): inclusion Criteria Single-segment Grade Ⅰ lumbar spondylolisthesis complicated with central spinal canal stenosis on imaging examinations; Accompanied by intermittent claudication, radiating pain and numbness of the lower extremities, and other relevant neurological symptoms; No relief of symptoms after more than 3 months of conservative treatment; The patient and their family members are fully informed of the trial details, have signed the informed consent form, and agree to participate in the trial.
  Exclusion Criteria Lumbar spondylolisthesis of Grade Ⅱ or higher; Non-degenerative lumbar spine diseases, or significant confirmed lumbar instability; Complicated with lumbar spine infection, tumor, trauma, or deformity; or with a history of previous lumbar spine surgery; Complicated with other systemic diseases that may significantly affect surgical efficacy (such as rheumatoid arthritis, severe osteoporosis, and severe mental illness).
  Interventions: Procedure: UBE
- PLIF/TLIF (Active Comparator): inclusion Criteria Single-segment Grade Ⅰ lumbar spondylolisthesis complicated with central spinal canal stenosis on imaging examinations; Accompanied by intermittent claudication, radiating pain and numbness of the lower extremities, and other relevant neurological symptoms; No relief of symptoms after more than 3 months of conservative treatment; The patient and their family members are fully informed of the trial details, have signed the informed consent form, and agree to participate in the trial.
  Exclusion Criteria Lumbar spondylolisthesis of Grade Ⅱ or higher; Non-degenerative lumbar spine diseases, or significant confirmed lumbar instability; Complicated with lumbar spine infection, tumor, trauma, or deformity; or with a history of previous lumbar spine surgery; Complicated with other systemic diseases that may significantly affect surgical efficacy (such as rheumatoid arthritis, severe osteoporosis, and severe mental illness).
  Interventions: Procedure: PLIF

INTERVENTIONS:
Procedure: UBE — Unilateral Biportal Endoscopy (UBE) for the treatment of lumbar spinal stenosis combines the advantages of both open surgery and minimally invasive surgery: ① Minimal surgical trauma: Only two small incisions of 0.8 cm are required, resulting in minimal damage to the paraspinal muscles; ② Aqueous medium surgical field: Radiofrequency can be used for effective and precise hemostasis under endoscopy, which significantly reduces blood loss; ③ Endoscopic operation: The surgical field is magnified, allowing clear and adequate exposure of the dura mater and nerves to avoid injury to important structural tissues; ④ Precise decompression: Under the above conditions, traditional surgical instruments and specialized tools such as endoscopic drills can be used to complete bilateral resection of the lamina and ligamentum flavum as well as spinal canal enlargement, achieving meticulous decompression of the central canal and lateral recess.
  Arms: Perform surgery using the Unilateral Biportal Endoscopy (UBE) technique
Procedure: PLIF — Posterior Lumbar Interbody Fusion (PLIF) adopts a midline posterior lumbar approach. On the basis of completing decompression of the spinal canal and nerve root canal, it resects the intervertebral disc tissue of the pathological segment and implants bone grafts (or interbody fusion cages) to achieve intervertebral bony fusion. Meanwhile, it is combined with a pedicle screw internal fixation system to maintain spinal alignment and stability, ultimately aiming to relieve neurological symptoms and restore the mechanical function of the spine.
  Arms: PLIF/TLIF

SUMMARY:
The research objective of this project is to clarify and compare the efficacy of the unilateral biportal endoscopy (UBE) technique and traditional open decompression, fusion and internal fixation surgery in the treatment of patients with Grade Ⅰ degenerative spondylolisthesis complicated with central spinal canal stenosis through high-quality, prospective, multicenter randomized controlled trials (RCTs), so as to provide high-level clinical research evidence for the expansion of UBE technique indications and its technical promotion.

DETAILED DESCRIPTION:
The selection of treatment methods for degenerative Grade Ⅰ spondylolisthesis complicated with lumbar spinal stenosis remains one of the controversial issues in the field of spinal surgery. Degenerative lumbar spondylolisthesis is a spinal sequence disorder caused by factors such as intervertebral disc degeneration and facet joint degeneration, with degeneration recognized as the primary driver of its onset and progression[1]. According to the Meyerding Classification, the severity of lumbar spondylolisthesis can be graded from Ⅰ to Ⅴ[2]. For spondylolisthesis of Grade Ⅱ or above accompanied by neurological symptoms, fusion and internal fixation surgery is generally indicated. In contrast, the surgical management of Grade Ⅰ spondylolisthesis with central spinal canal stenosis involves numerous clinically available approaches, including traditional open fusion surgery, minimally invasive techniques such as MIS-TLIF (Minimally Invasive Transforaminal Lumbar Interbody Fusion), OLIF (Oblique Lumbar Interbody Fusion), and spinal endoscopic surgery, all of which remain subject to ongoing debate[3]. Neither the 2011 Clinical Practice Guidelines for Degenerative Lumbar Spinal Stenosis issued by the North American Spine Society[4], the 2014 Chinese Expert Consensus on the Surgical Treatment Standards for Lumbar Spinal Stenosis[5], nor the 2023 Chinese Expert Consensus on the Diagnosis and Treatment of Degenerative Lumbar Spinal Stenosis[6] provides clear recommendations for the surgical treatment of Grade Ⅰ spondylolisthesis complicated with central spinal canal stenosis.

Unilateral Biportal Endoscopy (UBE)[7] is one of the most rapidly evolving technologies in spinal surgery in recent years, hailed as a minimally invasive spinal endoscopic technique "born for spinal stenosis". It can be applied to treat various lumbar degenerative diseases, including lumbar disc herniation and lumbar spinal stenosis. UBE employs two separate portals (one for endoscopic visualization and one for surgical manipulation) to perform minimally invasive procedures in coordination. As UBE is not restricted by instrument size, it is currently the most efficient among all minimally invasive spinal technologies. UBE for lumbar spinal stenosis integrates the advantages of both open and minimally invasive surgeries: ① Minimal surgical trauma, requiring only two small incisions of 0.8 cm each, with negligible damage to paraspinal muscles; ② Aqueous medium-based surgical field, allowing for effective and precise hemostasis using radiofrequency under endoscopic guidance, which significantly reduces blood loss; ③ Magnified endoscopic visualization enables clear and adequate exposure of the dura mater and nerves, avoiding injury to critical anatomical structures[8]; ④ Under the aforementioned conditions, traditional surgical instruments and specialized tools such as endoscopic drills can be used to achieve bilateral resection of the lamina and ligamentum flavum, as well as spinal canal enlargement, realizing meticulous decompression of the central canal and lateral recess[9]; ⑤ Patients can ambulate on the second day after surgery, with significantly reduced hospital stay, recovery time, postoperative pain, surgical infection rate, and intraoperative blood loss compared with other surgical modalities.

Currently, there is a paucity of international comparative studies between UBE and traditional lumbar spine surgeries. Some scholars have demonstrated through single-center, retrospective studies that compared with transforaminal endoscopic techniques, patients achieve significant improvements in postoperative VAS (Visual Analog Scale) and ODI (Oswestry Disability Index) scores, with the UBE group showing superior VAS and ODI scores within 6 months postoperatively, suggesting the therapeutic advantages of UBE[10]. Additionally, Tan et al. found that compared with traditional open surgery, patients with lumbar spinal stenosis who underwent UBE had shorter operation time, less intraoperative blood loss, shorter hospital stay, milder paraspinal muscle atrophy at 1 year postoperatively, and comparable clinical efficacy (assessed by SF-36, RNS, and RMDQ)[11], highlighting the advantages of UBE over traditional open lumbar spine surgery.

The applicant of this project has previously performed hundreds of UBE procedures. Based on the applicant's clinical experience and the summarized experiences of domestic and international scholars, UBE offers numerous benefits in the treatment of lumbar spinal stenosis. However, there remains significant controversy regarding the suitability of UBE for treating lumbar spinal stenosis complicated with degenerative Grade Ⅰ spondylolisthesis. The traditional viewpoint holds that due to the presence of spinal instability in Grade Ⅰ degenerative spondylolisthesis, simple decompression alone (without fusion) may fail to address the spondylolisthesis, necessitating decompression, reduction, fusion, and fixation to prevent progression of slippage, recurrence of neurological symptoms, and suboptimal clinical outcomes. From the perspective of minimally invasive surgery, the primary pathological issue in lumbar spinal stenosis with Grade Ⅰ degenerative spondylolisthesis is neurological compression caused by spinal stenosis; thus, relieving neurological compression via minimally invasive decompression alone can resolve patients' symptoms. This approach avoids complications associated with decompression plus internal fixation, such as nonunion, infection, and internal fixation failure. Furthermore, UBE causes minimal dissection of paraspinal muscles and negligible damage to facet joints, resulting in minimal impact on spinal stability and a low incidence of postoperative slippage progression or the need for reoperation with internal fixation. Nevertheless, there are currently no long-term clinical follow-up reports on UBE for lumbar spinal stenosis with Grade Ⅰ degenerative spondylolisthesis at home or abroad, and high-quality clinical evidence is particularly lacking.

The significance of this study lies in conducting a multicenter, prospective randomized controlled trial to comprehensively evaluate and compare the clinical efficacy, surgical complications, and postoperative quality of life between UBE and traditional open surgery for Grade Ⅰ degenerative spondylolisthesis complicated with lumbar spinal stenosis from multiple dimensions. This study aims to provide high-level clinical evidence for expanding the indications of UBE in minimally invasive spinal surgery and is expected to update or modify existing guidelines or expert consensus on the diagnosis and treatment of lumbar spinal stenosis.

Main Research Objectives To clarify the efficacy of the Unilateral Biportal Endoscopy (UBE) technique in the treatment of Grade Ⅰ degenerative spondylolisthesis complicated with central spinal canal stenosis; To compare the clinical outcomes between the UBE technique and traditional open decompression, fusion and internal fixation surgery; To provide high-level clinical research evidence for the expansion of UBE technique indications and its technical promotion.

ELIGIBILITY:
Inclusion Criteria Imaging findings: Single-segment Grade Ⅰ lumbar spondylolisthesis complicated with central spinal canal stenosis on imaging examinations; Clinical manifestations: Accompanied by intermittent claudication, radiating pain and numbness of the lower extremities, and other relevant neurological symptoms; Treatment history: No relief of symptoms after more than 3 months of conservative treatment; Informed consent: The patient and their family members are fully informed of the trial details, have signed the informed consent form, and agree to participate in the trial.

Exclusion Criteria Severe spondylolisthesis: Lumbar spondylolisthesis of Grade Ⅱ or higher; Non-degenerative or unstable conditions: Non-degenerative lumbar spine diseases, or significant confirmed lumbar instability; Special pathological or surgical history: Complicated with lumbar spine infection, tumor, trauma, or deformity; or with a history of previous lumbar spine surgery; Systemic comorbidities: Complicated with other systemic diseases that may significantly affect surgical efficacy (such as rheumatoid arthritis, severe osteoporosis, and severe mental illness).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
VAS | 24 months after surgery
  Status of Visual Analog Scale (VAS) Scores in Two Groups of Patients at 24 Months Postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No